CLINICAL TRIAL: NCT01986491
Title: An Open-Label, Single Dose, Relative Bioavailability Study of Solid Formulations in Fed and Fasted Conditions Followed by a Repeated Dose Study of a Selected Solid Formulation of JNJ-39393406 in Healthy Male Subjects
Brief Title: A Study of Solid Formulations of JNJ-39393406 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR016264; 39393406EDI1003 (Other: Johnson & Johnson Pharmaceutical Research & Development)
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Healthy
Keywords: Healthy; JNJ-39393406; Relative Bioavailability; Solid Formulation
MeSH Terms: interventions — Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Part 1; Period 1 (Experimental): Three participants will receive JNJ 39393406 of 2 different solid formulations (X and Y) with 2 different doses (30 mg and 120 mg) in following sequence (on Day 1 of each sequence) with a washout period of 1-2 weeks. 30 mg of solid X, 120 mg of solid Y, 30 mg of solid Y, and 120 mg of solid X.
  Interventions: Drug: JNJ 39393406 30 mg solid X; Drug: JNJ 39393406 30 mg solid Y; Drug: JNJ 39393406 120 mg solid X; Drug: JNJ 39393406 120 mg solid Y
- Part 1; Period 2 (Experimental): Three participants will receive JNJ 39393406 of 2 different solid formulations (X and Y) with 2 different doses (30 mg and 120 mg) in following sequence (on Day 1 of each sequence) with a washout period of 1-2 weeks. 30 mg of solid Y, 30 mg of solid X, 120 mg of solid X and 120 mg of solid Y.
  Interventions: Drug: JNJ 39393406 30 mg solid X; Drug: JNJ 39393406 30 mg solid Y; Drug: JNJ 39393406 120 mg solid X; Drug: JNJ 39393406 120 mg solid Y
- Part 1; Period 3 (Experimental): Three participants will receive JNJ 39393406 of 2 different solid formulations (X and Y) with 2 different doses (30 mg and 120 mg) in following sequence (on Day 1 of each sequence) with a washout period of 1-2 weeks: 120 mg of solid X, 30 mg of solid Y, 120 mg of solid Y, and 30 mg of solid X.
  Interventions: Drug: JNJ 39393406 30 mg solid X; Drug: JNJ 39393406 30 mg solid Y; Drug: JNJ 39393406 120 mg solid X; Drug: JNJ 39393406 120 mg solid Y
- Part 1; Period 4 (Experimental): Three participants will receive JNJ 39393406 of 2 different solid formulations (X and Y) with 2 different doses (30 mg and 120 mg) in following sequence (on Day 1 of each sequence) with a washout period of 1-2 weeks: 120 mg of solid Y, 120 mg of solid X, 30 mg of solid X, and 30 mg of solid Y.
  Interventions: Drug: JNJ 39393406 30 mg solid X; Drug: JNJ 39393406 30 mg solid Y; Drug: JNJ 39393406 120 mg solid X; Drug: JNJ 39393406 120 mg solid Y
- Part 2; Period 1 (Experimental): Four participants will receive 30 mg of JNJ 39393406 of 2 different formulations (solid formulation selected from Part 1 and solution) in following sequence (on Day 1 of each sequence) with a washout period of 1-2 weeks: 30 mg of solid formulation, and 30 mg of solution.
  Interventions: Drug: JNJ 39393406 30 mg solid X; Drug: JNJ 39393406 30 mg solid Y; Drug: JNJ 39393406 120 mg solid X; Drug: JNJ 39393406 120 mg solid Y; Drug: JNJ 39393406 30 mg solution
- Part 2; Period 2 (Experimental): Four participants will receive 30 mg of JNJ 39393406 of 2 different formulations (solid formulation selected from Part 1 and solution) in following sequence (on Day 1 of each sequence) with a washout period of 1-2 weeks: 30 mg of solution, and 30 mg of solid formulation.
  Interventions: Drug: JNJ 39393406 30 mg solid X; Drug: JNJ 39393406 30 mg solid Y; Drug: JNJ 39393406 120 mg solid X; Drug: JNJ 39393406 120 mg solid Y; Drug: JNJ 39393406 30 mg solution
- Part 3 (Experimental): Eight participants (same participants from Part 2) will receive JNJ 39393406 (dose will likely be 30 mg, or another multiple of the 30 mg solid dose form selected in Part 1, but not higher than 210 mg) from Days 1 to 7.
  Interventions: Drug: JNJ 39393406 30 mg solid X; Drug: JNJ 39393406 30 mg solid Y

INTERVENTIONS:
Drug: JNJ 39393406 30 mg solid X — Participants will receive JNJ 39393406 30 mg solid X formulation as a tablet orally (by mouth).
Drug: JNJ 39393406 30 mg solid Y — Participants will receive JNJ 39393406 30 mg solid Y formulation as a hard gelatin capsule orally (by mouth).
Drug: JNJ 39393406 120 mg solid X — Participants will receive JNJ 39393406 120 mg solid X formulation as a tablet orally (by mouth).
  Arms: Part 1; Period 1; Part 1; Period 2; Part 1; Period 3; Part 1; Period 4; Part 2; Period 1; Part 2; Period 2
Drug: JNJ 39393406 120 mg solid Y — Participants will receive JNJ 39393406 120 mg solid Y formulation as a hard gelatin capsule orally (by mouth).
  Arms: Part 1; Period 1; Part 1; Period 2; Part 1; Period 3; Part 1; Period 4; Part 2; Period 1; Part 2; Period 2
Drug: JNJ 39393406 30 mg solution — Participants will receive JNJ 39393406 30 mg/mL solution orally (by mouth).
  Arms: Part 2; Period 1; Part 2; Period 2

SUMMARY:
The purpose of the study is to compare the pharmacokinetics (what a medication does to the body), dose-proportionality, safety and tolerability of JNJ 39393406 following single dose oral administration of two solid oral formulations in Part 1; based on the profile in Part 1, one of the formulations assessed will be selected to investigate the pharmacokinetics in fasting condition in Part 2 and after repeated dosing in Part 3.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention) and single center study that will be conducted in 3 parts (Part 1, Part 2, and Part 3). The study consists of 3 phases including, the screening phase, treatment phase, and the follow-up phase. Part 1 is a four-way cross-over (method used to switch participants from one treatment arm to another in a clinical study) study to compare the pharmacokinetics, dose-proportionality, safety and tolerability of JNJ 39393406 following single dose oral administration of two solid oral formulations (X and Y). Approximately 12 participants will be enrolled in Part 1. Part 2 is two-way cross-over study in a separate group of participants to assess pharmacokinetics in fasting condition and the relative bioavailability (the extent to which a medication or other substance becomes available to the body) of the selected solid formulation from Part 1 compared with a solution formulation. Approximately 8 participants will be enrolled in Part 2. In Part 3, the single and repeated dose pharmacokinetics after administration of the selected formulation from Part 1 will be assessed for 7 consecutive days. The same participants will participate in Parts 2 and 3 of the study. Safety will be evaluated by the assessment of adverse events, clinical laboratory tests, electrocardiogram, vital signs, physical examination, and neurological examination. The duration of participation in the study for an individual participant will be approximately 8 weeks (including screening and follow up visit).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants
* Body mass index (BMI) between 18 and 30 kg/m2 (BMI is calculated as weight [kilogram] divided by square of height [meter])
* Willing to adhere to the prohibitions and restrictions specified in the protocol
* Must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Clinically significant abnormal values for clinical chemistry, hematology or urinalysis at screening or admission
* Clinically significant abnormal physical examination, neurological examination, vital signs or 12 lead electrocardiogram at screening
* Significant history of or current significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematological disease, bronchospastic respiratory disease, dyspnea, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, infection, or any other illness that the investigator considers clinically significant
* Significant history of or current psychiatric or neurological illness
* Serology positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus antibodies at screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration of JNJ 39393406 | Predose to 96 hrs postdose (Part 1 and Part 2 [after each single-dose administration]); predose to 24 hrs postdose (Day 1); predose to 5 hrs postdose (Days 3 and 5); predose to 96 hrs (Day 8), and end of study (7 to 14 days after the last dose) (Part 3)
  Maximum plasma concentration of JNJ 39393406, determined by visual inspection of the data
Time to reach the maximum plasma concentration of JNJ 39393406 | Predose to 96 hrs postdose (Part 1 and Part 2 [after each single-dose administration]); predose to 24 hrs postdose (Day 1); predose to 5 hrs postdose (Days 3 and 5); predose to 96 hrs (Day 8), and end of study (7 to 14 days after the last dose) (Part 3)
  Time to reach the maximum plasma concentration, determined by visual inspection of the data
Area under the plasma concentration-time curve of JNJ-39393406 | Predose to 96 hrs postdose (Part 1 and Part 2 [after each single-dose administration]); predose to 24 hrs postdose (Day 1); predose to 5 hrs postdose (Days 3 and 5); predose to 96 hrs (Day 8), and end of study (7 to 14 days after the last dose) (Part 3
Number of participants with adverse events | Up to 7 to 14 days after last dose of study medication (Part 1, Part 2, and Part 3)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Antwerp, Belgium